CLINICAL TRIAL: NCT03348969
Title: Neoadjuvant Short-term Intensive Chemoresection Versus Standard Adjuvant Intravesical Instillations in NMIBC
Acronym: NICSA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jørgen Bjerggaard Jensen (Other)
Responsible Party: Sponsor-Investigator, Jørgen Bjerggaard Jensen, Professor, MD, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DaBlaCa13
Record Dates: First submitted 2017-11-13; First posted 2017-11-21 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Bladder Cancer
Keywords: Mitomycin C; Neoadjuvant
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Mitomycin

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Neoadjuvant Mitomycin C
  Interventions: Drug: Mitomycin c
- Control (Active Comparator): Adjuvant Mitomycin C
  Interventions: Drug: Mitomycin c

INTERVENTIONS:
Drug: Mitomycin c — Neoadjuvant Mitomycin C
  Other Names: Mitomycin "Medac"

SUMMARY:
A randomized controlled trial aiming to investigate neoadjuvant, short-term intensive chemoresection with Mitomycin C compared to standard treatment with TURB and adjuvant intravesical instillation therapy in patients with recurrent non-muscle invasive bladder cancer (NMIBC).

DETAILED DESCRIPTION:
Background:

Bladder cancer is the 11th most common cancer in the world and one of the most costly cancers on a per patient basis, due to the cost of operative procedures, follow-up cystoscopies and instillation therapy. Furthermore there is a risk of progression to invasive and hence deadly cancer why efficient and immediate treatment is crucial. Treatment today consists of surgical removal of tumours (TURB) and adjuvant intravesical treatment. There is a chance; neoadjuvant intravesical treatment with chemotherapy can supersede surgical removal in chemo-sensitive tumours while however some tumours will not respond to intravesical chemotherapy. Currently it is not possible to predict which tumours are chemo-sensitive and which are not.

Objectives:

To assess the efficacy of neoadjuvant, short-term intensive chemoresection with Mitomycin C compared to standard treatment with TURB and adjuvant intravesical instillation therapy in patients with recurrent non-muscle invasive bladder cancer (NMIBC).

To investigate the ability to predict chemo-response in patients with recurrent non-muscle invasive bladder cancer (NMIBC).

Methods:

A randomised clinical controlled trial will include 120 patients with recurrent NMIBC.

The control group of 60 patients will receive standard care with TURB and adjuvant intravesical treatment. The intervention group of 60 patients will be submitted to neoadjuvant short-term intensive chemoresection with three instillations with Mitomycin C per week for two weeks. Remnant tumour tissue will be evaluated by flexible cystoscopy after four weeks.

To investigate the ability to predict chemo-response in patients with recurrent NMIBC, a connection between biomarkers of the initial tumour tissue and tumour response will be assessed.

Samples of the latest resected tumour prior to inclusion will be collected from all participants treated with neoadjuvant chemoresection and assessed against the tumour response seen in the trial.

Perspectives:

Validation of biomarkers to predict chemo-response will be an important step to integrate biomarkers in daily clinical practice and to individualize the treatment of NMIBC.

In some cases surgery could be avoided while ineffective chemotherapy could be avoided in others.

ELIGIBILITY:
Inclusion Criteria:

* Known history of urothelial non-invasive Ta-tumour low-grade or high-grade.
* ≥18 years old
* Mentally healthy individual
* The ability to understand Danish orally and in writing

Exclusion Criteria:

* Known history of invasive tumour of the bladder (T1+)
* Known history of CIS of the bladder
* Previous BCG-treatment within the last 24 months
* Previous Mitomycin C-treatment (except single-shot postoperative instillation)
* Known allergy or intolerance to Mitomycin C
* Solid tumour with suspicions of invasion
* Single tumour of more than 2 cm in diameter
* Suspicion of CIS (positive cytology with high-grade neoplastic cells combined with suspicious cystoscopy for flat lesions).
* Small bladder volume (less than 100 ml) or incontinence
* Acute cystitis
* Pregnancy or breast-feeding
* Not willing to use secure contraception with regard to men with partners and premenopausal women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year recurrence rate | within 2 years
  The primary outcome is the number of patients in need for a TURB or tumour fulguration in the first 2 years following randomization.
  TURBs included as primary endpoint are the initial TURB in the control group, the prospective TURB in the intervention group for patients without complete chemoresection as well as TURB due to recurrence in both study groups. In case a TURB is recommended, but a subject refuses to undergo surgery, the recommended TURB is also registered.

SECONDARY OUTCOMES:
Tumour response rate | 6 months after complete enrollment
  Number of patients with complete, partial and incomplete tumour response on neoadjuvant, short-term intensive chemoresection with Mitomycin C.
5-year recurrence rate | within 5 years
  The number of patients in need of a TURB or tumour fulguration in the outpatient clinic in the first 5 years following randomization.
  TURBs included are the initial TURB in the control group, the prospective TURB in the intervention group for patients without complete chemoresection as well as TURB due to recurrence in both study groups. In case a TURB is recommended, but a subject refuses to undergo surgery, the recommended TURB is also registered.
Adverse events | 6 months after complete enrollment
  Proportion of patients with adverse events related to neoadjuvant, short-term intensive chemoresection
Biomarkers | within 2 years
  Composition of 650 cancer-associated genes expressed on the last resected tumour

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen Bjerggaard Jensen, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herr H. Re: Marko Babjuk, Andreas Bohle, Maximilian Burger, et al. EAU Guidelines on Non-muscle-invasive Urothelial Carcinoma of the Bladder: Update 2016. Eur Urol 2017;71:447-61. Eur Urol. 2017 Jun;71(6):e171-e172. doi: 10.1016/j.eururo.2016.11.030. Epub 2016 Dec 12. No abstract available. PMID 27979427
- [Background] Maffezzini M. Re: Richard J. Sylvester, Adrian P.M. van der Meijden, Willem Oosterlinck, J. Alfred Witjes, Christian Bouffioux, Louis Denis and Donald W.W. Newling. Predicting recurrence and progression in individual patients with stage Ta T1 bladder cancer using EORTC risk tables: a combined analysis of 2596 patients from seven EORTC trials. Eur Urol 2006;49:466-77. Eur Urol. 2006 Sep;50(3):623-4; author reply 624-5. doi: 10.1016/j.eururo.2006.04.005. Epub 2006 May 4. No abstract available. PMID 16707208
- [Background] Kaasinen E, Wijkstrom H, Rintala E, Mestad O, Jahnson S, Malmstrom PU. Seventeen-year follow-up of the prospective randomized Nordic CIS study: BCG monotherapy versus alternating therapy with mitomycin C and BCG in patients with carcinoma in situ of the urinary bladder. Scand J Urol. 2016 Oct;50(5):360-8. doi: 10.1080/21681805.2016.1210672. Epub 2016 Aug 15. PMID 27603424
- [Background] Lamm DL. Preventing progression and improving survival with BCG maintenance. Eur Urol. 2000;37 Suppl 1:9-15. doi: 10.1159/000052376. PMID 10575266
- [Background] Shelley MD, Wilt TJ, Court J, Coles B, Kynaston H, Mason MD. Intravesical bacillus Calmette-Guerin is superior to mitomycin C in reducing tumour recurrence in high-risk superficial bladder cancer: a meta-analysis of randomized trials. BJU Int. 2004 Mar;93(4):485-90. doi: 10.1111/j.1464-410x.2003.04655.x. PMID 15008714
- [Background] Shida K, Shimasaki J, Takahashi H, Kurihara H, Sato J. [Therapy and prognosis of bladder tumors--result of injection of mitomycin C into the bladder]. Gan No Rinsho. 1970 Jul;16(7):737-44. No abstract available. Japanese. PMID 5465489
- [Background] Colombo R, Rocchini L, Suardi N, Benigni F, Colciago G, Bettiga A, Pellucchi F, Maccagnano C, Briganti A, Salonia A, Rigatti P, Montorsi F. Neoadjuvant short-term intensive intravesical mitomycin C regimen compared with weekly schedule for low-grade recurrent non-muscle-invasive bladder cancer: preliminary results of a randomised phase 2 study. Eur Urol. 2012 Nov;62(5):797-802. doi: 10.1016/j.eururo.2012.05.032. Epub 2012 May 18. PMID 22633362
- [Background] Sousa A, Inman BA, Pineiro I, Monserrat V, Perez A, Aparici V, Gomez I, Neira P, Uribarri C. A clinical trial of neoadjuvant hyperthermic intravesical chemotherapy (HIVEC) for treating intermediate and high-risk non-muscle invasive bladder cancer. Int J Hyperthermia. 2014 May;30(3):166-70. doi: 10.3109/02656736.2014.900194. Epub 2014 Apr 3. PMID 24697672
- [Background] Miyata Y, Sakai H. Predictive Markers for the Recurrence of Nonmuscle Invasive Bladder Cancer Treated with Intravesical Therapy. Dis Markers. 2015;2015:857416. doi: 10.1155/2015/857416. Epub 2015 Nov 23. PMID 26681820
- [Background] Seo HK, Cho KS, Chung J, Joung JY, Park WS, Chung MK, Lee KH. Prognostic value of p53 and Ki-67 expression in intermediate-risk patients with nonmuscle-invasive bladder cancer receiving adjuvant intravesical mitomycin C therapy. Urology. 2010 Aug;76(2):512.e1-7. doi: 10.1016/j.urology.2010.04.040. Epub 2010 Jun 26. PMID 20579709
- [Background] Chen JX, Deng N, Chen X, Chen LW, Qiu SP, Li XF, Li JP. A novel molecular grading model: combination of Ki67 and VEGF in predicting tumor recurrence and progression in non-invasive urothelial bladder cancer. Asian Pac J Cancer Prev. 2012;13(5):2229-34. doi: 10.7314/apjcp.2012.13.5.2229. PMID 22901199
- [Background] Karam JA, Lotan Y, Ashfaq R, Sagalowsky AI, Shariat SF. Survivin expression in patients with non-muscle-invasive urothelial cell carcinoma of the bladder. Urology. 2007 Sep;70(3):482-6. doi: 10.1016/j.urology.2007.05.009. PMID 17905101
- [Background] Bracci L, Schiavoni G, Sistigu A, Belardelli F. Immune-based mechanisms of cytotoxic chemotherapy: implications for the design of novel and rationale-based combined treatments against cancer. Cell Death Differ. 2014 Jan;21(1):15-25. doi: 10.1038/cdd.2013.67. Epub 2013 Jun 21. PMID 23787994
- [Background] Hugo W, Zaretsky JM, Sun L, Song C, Moreno BH, Hu-Lieskovan S, Berent-Maoz B, Pang J, Chmielowski B, Cherry G, Seja E, Lomeli S, Kong X, Kelley MC, Sosman JA, Johnson DB, Ribas A, Lo RS. Genomic and Transcriptomic Features of Response to Anti-PD-1 Therapy in Metastatic Melanoma. Cell. 2017 Jan 26;168(3):542. doi: 10.1016/j.cell.2017.01.010. No abstract available. PMID 28129544
- [Derived] Lindgren MS, Hansen E, Azawi N, Nielsen AM, Dyrskjot L, Jensen JB. DaBlaCa-13 Study: Oncological Outcome of Short-Term, Intensive Chemoresection With Mitomycin in Nonmuscle Invasive Bladder Cancer: Primary Outcome of a Randomized Controlled Trial. J Clin Oncol. 2023 Jan 10;41(2):206-211. doi: 10.1200/JCO.22.00470. Epub 2022 Oct 12. PMID 36223555